CLINICAL TRIAL: NCT00361426
Title: EarlySense Monitoring Device Evaluation on Patients in Med / Surg
Brief Title: EarlySense Monitoring Device Evaluation on COPD, CHF and Pneumonia Patients
Status: Withdrawn | Type: Observational
Why Stopped: No need
Sponsor: EarlySense Ltd. (Industry)
Collaborators: The Chaim Sheba Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 022-05B
Record Dates: First submitted 2006-08-06; First posted 2006-08-08 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2008-01

CONDITIONS: COPD Patients
Keywords: COPD; Respiration Rate; Monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Earlysense vital sign monitor — The system is a contactless system that measures heart and respiratory rates and other parameters via a contactless sensor that is placed under the patient mattress
  Other Names: EarlySense system device

SUMMARY:
Continuous measurement of breathing patterns, heart rate, restlessness and cough in sleep using EarlySense ES 16 device. Predicting worsening in COPD patients' condition using the above parameters.

DETAILED DESCRIPTION:
Study's participants are CHF, COPD and Pneumonia patients or patients who are otherwise hospitalized in internal medicine department. During the study the patients' breathing patterns, heart rate, restlessness and cough in sleep will be measured by the EarlySense ES 16 device, which is placed in the patients' bed.

Patients' clinical status are followed. The patient's clinical condition is followed and analyzed in comparison to the EarlySense system output in order to determine the capability of the EarlySense system to predict COPD, CHF or Pneumonia deteriorations.

ELIGIBILITY:
Inclusion Criteria:

* CHF, COPD and Pneumonia Patients or control group non respiratory patients
* 18 years old and up
* Able to perform spirometry test or connect to ECG, respiratory belt, SPO2
* Willing to sign consent form
* Home close to Tel Aviv

Exclusion Criteria:

* hospitalization within the passing year

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in Med/Surg unit
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martine Szyper-Kravitz, M.D., Principal Investigator — Haim Sheba Medical Center, Israel
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel